CLINICAL TRIAL: NCT04033211
Title: Randomized, Multi-center, Double Blinded, Prospective Study to Evaluate the Incidence of Complications in Laparoscopic Cholecystectomy and Appendectomy Using Novosyn® CHD Versus Novosyn® Suture Material to Close Trocar Wound
Brief Title: NOVOsyn® for Trocar Incision After Laparoscopic Appendectomy and Cholecystectomy
Acronym: NOVOTILAC
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1816
Record Dates: First submitted 2019-07-04; First posted 2019-07-26 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Appendicitis; Cholecystitis
Keywords: Minimal invasive surgery; Appendectomy; Cholecystectomy
MeSH Terms: conditions — Appendicitis; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novosyn® CHD: A population undergoing a primary emergency or early elective (24h - 7 days) laparoscopic appendectomy or a primary emergency or early elective laparoscopic cholecystectomy using Novosyn® CHD suture for fascia and skin closure of trocar wounds.
  Interventions: Device: Novosyn® CHD for fascia and skin closure
- Novosyn®: A population undergoing a primary emergency or early elective (24h - 7 days) laparoscopic appendectomy or a primary emergency or early elective laparoscopic cholecystectomy using either Novosyn® suture for fascia and skin closure of trocar wounds.
  Interventions: Device: Novosyn® for fascia and skin closure

INTERVENTIONS:
Device: Novosyn® CHD for fascia and skin closure — Experimental
  Groups: Novosyn® CHD
Device: Novosyn® for fascia and skin closure — Comparator
  Groups: Novosyn®

SUMMARY:
The aim of this study is to evaluate if the application of a Chlorhexidine coated suture (Novosyn® CHD) will reduce the colonization of bacteria in comparison to an uncoated suture (Novosyn®) used for the closure of trocar wounds in laparoscopic surgery (appendectomy and cholecystectomy).

DETAILED DESCRIPTION:
The bacteriostatic and bactericidal effect of Novosyn® CHD will be assessed by the incidence of surgical site infection (SSI) in each suture group until 30 days postoperatively. The frequency of infections (SSI: A1 and A2) is considered as a suitable parameter for the assessment of efficacy. It is expected that the use of the Novosyn® CHD suture will reduce the occurrence of infections (SSI: A1 and A2) 30 days postoperatively compared to Novosyn suture (primary objective). SSI will be classified according to the Centre of Disease Control and Prevention (CDC), therefore the time point for assessment of SSI as set to 30 days postoperatively.

Furthermore, short-term and long-term complications, the handling of the suture material, length of postoperative hospital stay, costs, pain, quality of life, time to return to work, hernia rate including umbilical hernias and the cosmetic outcome will also be assessed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary emergency or early elective (24h - 7 days) laparoscopic appendectomy or cholecystectomy.
* Written informed consent
* Age≥ 18 years
* Not incapacitated patient

Exclusion Criteria:

* Open surgery for appendectomy or cholecystectomy
* Pregnancy
* Allergy or hypersensitivity to chlorhexidine
* Intraoperatively conversion from laparoscopic to open surgery
* Patients taking medical consumption that might affect wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population undergoing a primary emergency or early elective (24h - 7 days) laparoscopic appendectomy or a primary emergency or early elective laparoscopic cholecystectomy using either Novosyn® CHD or Novosyn® suture for fascia and skin closure of trocar wounds.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | until 30 days + 10 days after surgery
  Incidence of postoperative surgical site infections, SSI (A1: Superficial incisional site infections and A2: Deep incisional surgical site infections) (efficacy parameter) Surgical Site Infection (SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC).

SECONDARY OUTCOMES:
Development of Wound Dehiscence | until discharge (ca. 10 days postop), 30 days +10 days and 1 year ±2 months postoperatively
  Incidence of wound dehiscence (skin) at different postoperative examinations
Reoperation Rate | until discharge (ca. 10 days postop), 30 days +10 days and 1 year ±2 months postoperatively
  Incidence of reoperation rate at different postoperative times
Mortality Rate | until discharge (ca. 10 days postop), 30 days +10 days, and 1 year ±2 months postoperatively
  Incidence of mortality rate at different postoperative times
Postoperative Complications during the postoperative Course | until discharge (ca. 10 days postop), 30 days +10 days, 1 year ±2 months postoperatively
  Rates of postoperative complications such as bleeding, tissue reaction, abscess, perforation, bile leaks, biliary peritonitis, ileus, stenosis, fistula at different postoperative points in time
Suture Removal due to Wound Problems during the postoperative Course | until discharge (ca. 10 days postop), 30 days +10 days, and 1 year ±2 months postoperatively
  Rate of suture removal due to wound problems (infection, dehiscence, residual material requiring removal) at different defined postoperative points in time
Length of hospital stay | until discharge (ca. 10 days postop)
  Defined as the time period from day of operation until day of discharge (efficacy parameter).
Postoperative Surgical Site Infections | 1 year ±2 months post-op
  Incidence of postoperative surgical site infections
Rate of Conversion to open surgery | intraoperatively
  Number of interventions where operation technique has to be converted to open surgery intraoperatively
Time to return to work | up to 1 year ±2 months
  Defined as the duration (days) from day of surgery until the day when the patient was able to work. Employment status of the patient will also be reported.
Course of Pain: Visual Analogue Scale (VAS) | preoperatively, at day of discharge (ca. 10 days postop), at 30 days +10 days and 1 year ±2 months postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain". The values are compared over postoperative period.
Course of Cosmetic result | 30 days +10 days, 1 year ±2 months postoperatively
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum)
Course of Overall patient and observer satisfaction with the scar: Patient and Observer Scar Assessment Scale (POSAS) | 30 days +10 day, 1 year ±2 months postoperatively
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum)
Comparison of wound appearance | discharge (ca. 10 days postop), 30 days +10 days and 1 year ±2 months postoperatively
  Photographic documentation of the wounds for assessment
Comparison of handling parameters of the suture materials | intraoperatively
  Comparison of the handling features of the suture materials in eight different categories (ease of passage of the suture, first throw knot holding, knot tie down smoothness, knot security, surgical hand, memory effect, lack of frying and the overall handling) by rating each category on a 5 point scale (excellent, very good, good, satisfied, poor); no overall score is calculated, the categories are compared separately
Course of Health Status | 30 days +10 days after surgery, 1 year ±2 months after surgery
  EQ-5D is a standardised measure of health status developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D is designed for self-completion by respondents and it takes only a few minutes to complete. Instructions to respondents are included in the questionnaire. EQ-5D-5L consists of 2 pages - descriptive system and the EQ visual Analogue scale (EQ-VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the respondents self rated health on a 20 cm vertical , visual analogue scale with endpoints labelled "the best health you can imagine" and " the worst health you can imagine"
Hernia Rate / Umbilical Hernia Rate | until discharge (ca. 10 days postop), 30 days +10 days, 1 year ±2 months postoperatively
  Hernia rate including umbilical hernia postoperatively verified by ultra-sound examination compared at different postoperative points in time
Costs (economics) | 1 year ±2 months
  Assessment of costs will be calculated on postoperative complication (SSI) in both suture groups (efficient parameter).

CONTACTS AND LOCATIONS:
Overall Officials: Markus Golling, Prof. Dr., Principal Investigator — Diakonie Klinikum gGmbH Schwäbisch Hall
Locations (4):
- Germany (2):
  - Klinikverbund Südwest Krankenhaus Leonberg Alllgemeinchirurgie, Leonberg, Baden-Wurttemberg
  - Diakonie Klinikum gGmbH Schwäbisch Hall, Schwäbisch Hall, Baden-Wurttemberg
- Spain (2):
  - Hospital Germans Trias i Pujol General and Digestive Surgery, Badalona
  - General Surgery Department Hospital Plató, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Golling MT, Breul V, Barongo S, Milosheski T, Rubio JC, Pinedo AZ, Hoyuela C, Hidalgo NJ, Steurer W, Baumann P. Chlorhexidine - coated vs non-coated Suture to prevent surgical site infections following laparoscopic abdominal surgery (a prospective, randomized, controlled trial; NOVOTILAC). Langenbecks Arch Surg. 2025 Jun 13;410(1):191. doi: 10.1007/s00423-025-03757-x. PMID 40512393
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/40512393/